CLINICAL TRIAL: NCT00636012
Title: Stimulation of Gastric Slow Waves by Acupuncture of St36 and Pe6 - a Randomized Single-blind Controlled Trial
Brief Title: Stimulation of Gastric Slow Waves With Acupuncture at St36 and Pe6 - a Randomized Single-blind Controlled Trial
Acronym: GSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia M. Witt, Prof. Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: GSW-08
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Acupuncture
Keywords: acupuncture; Acupuncture points

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): verum acupuncture
  Interventions: Procedure: verum acupuncture
- 2 (Sham Comparator): sham acupuncture
  Interventions: Procedure: sham acupuncture

INTERVENTIONS:
Procedure: verum acupuncture — acupuncture at St36 and Pe6
  Arms: 1
Procedure: sham acupuncture — superficial needling at sham points
  Arms: 2

SUMMARY:
Aim of the study is to investigate specific effects of acupuncture points.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* BMI between 17.5 and 25
* 3 hours before the experiment no food
* 3 hours before the experiment only water, and 1 hour before the experiment no fluid intake
* 4 hours before the experiment no smoking
* informed consent

Exclusion Criteria:

* acupuncture treatment during the last 12 months
* chronic disease
* regular intake of medication which influence autonomic nervous system or GI tract
* pregnant or breast feeding
* drug or substance abuse

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
increase of percentage of regular gastric slow waves in the acupuncture group compared to the control group | baseline, acupuncture

SECONDARY OUTCOMES:
increase of percentage of regular gastric slow waves in acupuncture with stimulation compared to no stimulation | baseline, acupuncture
half cycles | baseline, acupuncture
systolic blood pressure | baseline, acupuncture
diastolic blood pressure | baseline, acupuncture
mean blood pressure | baseline, acupuncture
variability of heart rate | baseline, acupuncture
heart rate | baseline, acupuncture
breathing rate | baseline, acupuncture
skin conductance level | baseline, acupuncture
total vascular resistance | baseline, acupuncture
stroke volume | baseline, acupuncture
correlation between percentage of regular gastric slow waves and secondary outcome measures | baseline, acupuncture
impact of needle sensation on gastric slow waves | baseline, acupuncture
impact of expectation on gastric slow waves | baseline, acupuncture
impact of anxiety (state-trait-anxiety-inventory) on gastric slow waves | baseline, acupuncture

CONTACTS AND LOCATIONS:
Overall Officials: Claudia M. Witt, MD, Principal Investigator — Institute for Social Medicine, Epidemiology, and Health Economics, Charité University Medical Center, Berlin, Germany; Frank Zimmermann-Viehoff, MD, Principal Investigator — Department Psychosomatics and Psychotherapy, Charité University Medical Center, Berlin, Germany
Locations (1):
- Charité University Medical Center, Berlin, Germany

REFERENCES:
- [Result] Witt CM, Meissner K, Pach D, Thiele C, Ludtke R, Ghadiyali Z, Deter HC, Zimmermann-Viehoff F. Stimulation of gastric slow waves with manual acupuncture at acupuncture points ST36 and PC6--a randomized single blind controlled trial. Neurogastroenterol Motil. 2012 May;24(5):438-45, e211-2. doi: 10.1111/j.1365-2982.2012.01877.x. Epub 2012 Feb 6. PMID 22309404